CLINICAL TRIAL: NCT06862323
Title: Does Timing Matter? A Trial of Time Restricted Eating in Haematological Malignancies
Brief Title: Time Restricted Eating in Haematological Malignancies
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: British Columbia Cancer Agency (Other)
Collaborators: BC Cancer Foundation (Other); Michael Smith Foundation for Health Research (Other)
Responsible Party: Principal Investigator, Eleah Stringer, Clinical and Research Dietitian, British Columbia Cancer Agency
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: H24-01236
Record Dates: First submitted 2025-03-03; First posted 2025-03-06 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Cancer; Chronic Lymphocytic Leukemia
Keywords: Time Restricted Eating; Intermittent Fasting; Diet; Cancer; Chronic Lymphocytic Leukemia; Autophagy; Microbiome; Inflammation; Epigenetics
MeSH Terms: conditions — Neoplasms; Leukemia, Lymphocytic, Chronic, B-Cell; Intermittent Fasting; Inflammation

STUDY DESIGN:
Intervention Model Description: A dietary intervention of intermittent fasting will be provided to the experimental arm of people with cancer and control arm of people without cancer.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Research Design: A nonrandomized control design will be followed with a 4:1 ratio (experimental: control). The experimental arm will consist of patients with early stage CLL who are on surveillance (n=60). Participants will follow a fasting intervention of an 8-hour feeding window with a 16-hour fasting window for a minimum of 6/7 days per week for either 3 months (90 days) or 6 months (180 days) based on their preference. Participants with cancer will provide blood samples, stool samples (optional) and will complete journals, check ins, and quality of life surveys per the schedule outlined in section 5.7 as well as in the attached study protocol document in section 6. Upon completion of study, participants with cancer may also complete an optional end of study interview.
  Interventions: Behavioral: Time-Restricted Eating
- Control Group (Active Comparator): The control arm will consist of community members who do not have cancer (n=15). Participants will follow a fasting intervention of an 8-hour feeding window with a 16-hour fasting window for a minimum of 6/7 days per week for either 3 months (90 days) or 6 months (180 days) based on their preference. Control participants will provide blood samples and weekly journals to serve as a control for autophagy flux analysis.
  Interventions: Behavioral: Time-Restricted Eating

INTERVENTIONS:
Behavioral: Time-Restricted Eating — TRE will be defined as a 16 hour fast with an 8 hour feeding window, with the option of a longer feeding window one day per week. All participants will adhere to the fasting intervention for either 90 days (3 months) or 180 days (6 months) based on their preference. Participants will be provided guidance (see appendix 7, Fasting Guidelines) on how to achieve an 8 hour feeding window by day 9 of the study and are recommended to adhere to the 16 hour fast/8 hour feeding window daily for the remainder of the study.

SUMMARY:
The goal of this clinical trial is to learn if time restricted eating (TRE), a form of intermittent fasting, can impact health outcomes in patients with chronic lymphocytic leukemia (CLL). The main questions it aims to answer are:

* In patients with CLL, is there a decrease or stabilization in cancer cell counts associated with TRE compared to baseline?
* Is there a decrease in immune cell autophagy (a cellular recycling process) activity associated with TRE compared to baseline?
* Does adherence to a TRE regimen improve patient experience and quality of life?

Immune cell autophagy activity in cancer patients will be compared to a subset of control participants without cancer.

Participants will:

* Adhere to a 16/8 fasting regimen, which involves eating as normal for 8 hours per day and fasting (only consuming water, black coffee or black tea) for the remaining 16 hours. They will follow this intervention for their choice of either 3 or 6 months.
* Complete monthly blood collections
* Complete weekly journal entries to record weekly weight and timing of first and last daily meals
* Complete weekly safety check-ins with a study team member for the first 4 weeks of the study and then bi-weekly thereafter
* Complete 3 quality of life questionnaires
* Provide 3 stool samples (optional component of study)
* Complete an end of study interview (optional component of study)

ELIGIBILITY:
Inclusion Criteria:

Experimental Participants:

* Diagnosis of CLL or SLL, Age 18-85
* Peripheral blood lymphocytes >20 x 10^9/L
* Hemoglobin >90g/L
* Platelets ˃90 x 10^9/L
* BMI of >=20kg/m2
* ECOG Performance Status >=2
* Not following any form of IF for 4 months prior to study

Control Participants:

* Absence of cancer diagnosis (active or historical)
* Age 18-85, Peripheral blood lymphocytes <5 x10^9/L
* BMI of >=20kg/m2
* ECOG Performance Status >=2
* Not following any form of IF for 4 months prior to study

Exclusion Criteria:

Experimental and Control Participants:

* Unable to give consent
* On medications required to be taken with food during the fasting window
* Pregnant or breastfeeding
* Diabetes mellitus
* BMI drop to < 18.5kg/m2 at any time during study
* Anti-lymphoma therapy within the past 3 months
* Expected to initiate anti-lymphoma therapy within the next 3 months
* Unable to fast due to a digestive system disorder
* > 85 years of age (due to frailty, increased risk of infection, and burden of additional blood collections)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Blood Sample Lymphocyte Count | 3 months
  Lymphocyte count assessment will be made at pre-intervention (within 3 months of the start of the IF study period), then monthly. If participants opt for a 90-day fast, blood collections will be completed on day 1, 30, 60, 90 and one month after completion of the TRE study period, to examine if TRE had an effect on lymphocyte numbers. Participants who opt for the 180-day fast will complete blood collections on day 1, 30, 60, 90, 120, 150 and 180. Blood collected at these time points will be analyzed for autophagy activation and for changes in immune, inflammatory, metabolic and epigenetic parameters.
Blood Sample Autophagy Flux Analysis | 3 months
  Participants will provide blood samples for autophagy flux analysis.
Epigenetic Analysis via PBMC Profiling | 3 months
  PBMC Profiling
Microbiome Analysis of Stool Samples | 3 months
  Optionally, stool samples will be collected for microbiome analysis.

SECONDARY OUTCOMES:
Participant Experience: QLQ-30 and FACITF Questionnaires | 3 months
  Descriptive statistics will characterize study participants and quality of life indicators from QLQ-30 and FACITF questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Eleah Stringer, MSc, RD, CSO, Principal Investigator — BC Cancer
Locations (1):
- BC Cancer, Victoria, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Yes
IPD will be available through OSF upon study completion. The protocol will be published.
Supporting Information: SAP, CSR, Analytic Code
Time Frame: Will be available upon study completion (estimated date of September 2027) and will remained available for 10 years.
Access Criteria: The aforementioned data will be made publicly available following study completion via OpenScienceFramework webpage. Additional data may be shared upon requested to study Principal Investigator.

REFERENCES:
- [Background] Stringer EJ, Cloke RWG, Van der Meer L, Murphy RA, Macpherson NA, Lum JJ. The Clinical Impact of Time-restricted Eating on Cancer: A Systematic Review. Nutr Rev. 2025 Jul 1;83(7):e1660-e1676. doi: 10.1093/nutrit/nuae105. PMID 39212676
- See also: Description of research program — https://www.bccrc.ca/dept/nahr/intermittent-fasting-oncology-studies-test